CLINICAL TRIAL: NCT06375707
Title: Efficacy and Safety of Ribociclib in Combination With NSAI Versus Physician's Choice of Chemotherapy Sequential Endocrine Therapy in HR+/HER2- Advanced Breast Cancer: a Phase II Randomised Controlled Clinical Trial
Brief Title: Efficacy and Safety of Ribociclib in Combination With NSAI Versus Physician's Choice of Chemotherapy Sequential Endocrine Therapy in HR+/HER2- Advanced Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HERO-KC23
Record Dates: First submitted 2023-12-28; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Advanced Breast Cancer
Keywords: HR positive /HER2 negative; Ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- physician's choice of chemotherapy sequential Ribociclib combined with NSAI±OFS (Active Comparator)
  Interventions: Drug: physician's choice of chemotherapy sequential Ribociclib combined with NSAI±OFS
- Ribociclib combined with NSAI±OFS (Experimental)
  Interventions: Drug: Ribociclib combined with NSAI±OFS

INTERVENTIONS:
Drug: physician's choice of chemotherapy sequential Ribociclib combined with NSAI±OFS — Docetaxel: 100mg/m2 IV every 21 days Paclitaxel: 175mg/m2 every 21 days, IV drip Vinorelbine: 25mg/ m2 on days 1 and 8 of each cycle, 1 cycle in 21 days, IV drip Capecitabine: 1000mg/m2, 2 times/d, 2 consecutive weeks of oral discontinuation for 1 week.
  Ribociclib: 600mg /d, 3 weeks continuous oral withdrawal for 1 week NSAI: Anastrozole 1mg, 1 time /d, oral or Letrozole: 2.5mg, 1 time /d, oral
  Arms: physician's choice of chemotherapy sequential Ribociclib combined with NSAI±OFS
Drug: Ribociclib combined with NSAI±OFS — Ribociclib: 600mg /d, 3 weeks continuous oral withdrawal for 1 week NSAI: Anastrozole 1mg, 1 time /d, oral or Letrozole: 2.5mg, 1 time /d, oral
  Arms: Ribociclib combined with NSAI±OFS

SUMMARY:
Evaluate the efficacy and safety of Ribociclib in combination with NSAI versus physician's choice of chemotherapy sequential endocrine therapy in HR+/HER2- advanced breast cancer.

DETAILED DESCRIPTION:
The main goal of this clinical trial is to compare in the efficacy of Ribociclib in combination with NSAI versus physician's choice of chemotherapy sequential endocrine therapy in HR+/HER2- advanced breast cancer and evaluate the PCR DFS,OS and safety of the subjects. The main question it aims is comparing the efficacy and safety of first-line application of CDK4/6 inhibitors combined with initial endocrine therapy versus sequential endocrine therapy after chemotherapy induction therapy in HR+/HER2-advanced breast cancer with rapidly progressive disease.

This study is planned to include 144 patients with HR+/HER2-advanced breast cancer with rapidly progressive disease between November 2023 and November 2025 who meet the entry criteria. A central dynamic randomisation system was used for 1:1 allocation to the repositories combined with NSAI treatment group and the physician's choice of chemotherapy sequential repositories combined with NSAI treatment group, with stratification factors including: level of HR expression, and presence of liver/lung metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is an adult female ≥ 18 years old at the time of informed consent.
2. ECGO rating 0-2.
3. Histologically confirmed recurrent or metastatic breast cancer, including patients initially diagnosed as stage IV or locally advanced inoperable patients.
4. Patient has a histologically and/or cytologically confirmed diagnosis of estrogen-receptor positive and/or progesterone receptor positive breast cancer based on the most recently analyzed tissue sample and all tested by local laboratory. ER should be more than 10% ER positive by local laboratory testing.
5. Patient has HER2-negative breast cancer defined as a negative in situ hybridization test or an IHC status of 0, 1 + or 2 + If IHC is 2 +, a negative in situ hybridization (FISH, CISH, or SISH) test is required by local laboratory testing and based on the most recently analyzed tissue sample.
6. Determination by the physician that the patient is in a rapid disease progression situation:

   * Symptomatic visceral metastases
   * Rapid progression of disease or impending visceral compromise.
   * Markedly symptomatic non visceral disease if the treating physician opt to give chemotherapy for rapid palliation of patients symptoms.
7. Patient hasn't received systemic anti-cancer therapy at the stage of recurrence/metastasis.
8. Patient must have at least one measurable lesion (according to RECIST 1.1 criteria)
9. Postmenopausal or pre/perimenopausal female patients are eligible for enrolment; pre or perimenopausal female patients must be willing to receive LHRHa during the study period.
10. All patients were required to meet the following laboratory biochemical values prior to enrolment:

    * Haematology: Hb ≥90 g/L, WBC ≥3.5×109/L, ANC ≥1.5×109/L, PLT ≥100×109/L;
    * Renal function: serum creatinine ≤ upper limit of normal value;
    * Liver function: for those without liver metastases, AST, ALT, ALP ≤2.5 times the upper limit of normal values, and ≤1.25 x the upper limit of normal values for total bilirubin; for those with liver metastases, AST, ALT, ALP ≤ 5 times the upper limit of normal value, and total bilirubin ≤ 1.5 x upper limit of normal value.

Exclusion Criteria:

1. Patient has received systemic anti-cancer therapy at the stage of recurrence/metastasis.
2. Those who have been treated with CDK4/6 inhibitors in the neoadjuvant/adjuvant phase.
3. Patients those with symptomatic CNS metastases.
4. Patient has a history of clinically symptomatic cardiovascular, hepatic, respiratory, renal and haemato-endocrine system or neuropsychiatric disorders.
5. Patient has a serious concomitant disease, such as an infectious disease; has multiple factors that affect the oral administration and absorption of the drug.
6. Pregnant or lactating women (women of childbearing age must have had a negative pregnancy test within 14 days prior to the first dose; if positive, pregnancy must be ruled out by ultrasound).
7. Patients in poor general condition who cannot tolerate chemotherapy treatment.
8. The investigator considers the patient unsuitable for entry into this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patient is an adult female ≥ 18 years old at the time of informed consent.
Enrollment: 144 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Progression-free survival is defined as the time from the date of randomization to the date of the first documented progression as per local review and according to RECIST 1.1 or death due to any cause.

SECONDARY OUTCOMES:
Progression Free Survival2 | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Refers to the time from randomization to disease progression or death after a patient enters a clinical trial and receives second-line therapy.
Time to treatment failure | From randomization to treatment failure or withdrawal from the trial; reasons for withdrawal can be patient request, disease progression, death, or adverse events, whichever came first, assessed up to 100 months
  Time to treatment failure is defined as the time from the date of randomization/start of treatment to the earliest of date of progression, date of death due to any cause, change to other anti-cancer therapy, or date of discontinuation due to reasons other than 'Protocol violation' or 'Administrative problems'.
Overall response rate (ORR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Overall response rate (ORR) is defined as the proportion of patients whose best overall response is either complete response (CR) or partial response (PR), as per local review and according to RECIST 1.1.
Overall survival(OS) | From date of randomization until the date of death from any cause, assessed up to 100 months
  Overall survival is defined as the time from the date of randomization to the date of death due to any cause.
Time To Response (TTR) | From the date of randomization to the first documented response of either CR or PR, whichever came first, assessed up to 100 months
  Time to response is defined as the time from the date of randomization to the first documented response of either CR or PR, which must be subsequently confirmed, as defined by RECIST 1.1.
Clinical benefit rate(CBR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Clinical benefit rate is defined as the proportion of patients with a best overall response of CR, or PR or stable disease, lasting for a duration of at least 24 weeks, as defined by RECIST 1.1.
Change from baseline in the global health status/QOL scale score by using FACT-B questionnaire | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Functional Assessment of Cancer Therapy - Breast (FACT-B) will be collected to assess health-related QoL, health status, functioning, disease symptoms, side effects, and cancer-related pain.
  Descriptive statistics will be used to summarize the overall score at each scheduled assessment time point. Additionally, change from baseline at the time of each assessment will be summarized.
  The distribution of time to definitive 10% deterioration in the global health status from FACT-B questionnaire will be assessed in the two treatment arms. Scores range from 0 to 4. no subscale. 0 score is the worst for social/family and functional wellbeing and 4 is the worst for physical, emotional wellbeing and additional concerns.
Frequency/severity of adverse events, lab abnormalities | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Safety of ribociclib in combination with NSAI and OFS, and combination chemotherapies

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial People's Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code